CLINICAL TRIAL: NCT07019038
Title: National Longitudinal Cohort of Hematological Diseases- Autoimmune Hemolytic Anemia
Acronym: NICHE-AIHA
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: IIT2025042
Record Dates: First submitted 2025-05-28; First posted 2025-06-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: AIHA - Warm Autoimmune Hemolytic Anemia; AIHA - Cold Autoimmune Hemolytic Anemia; Autoimmune Hemolytic Anemia Mixed Type
Keywords: Autoimmune Hemolytic Anemia; Treatment patterns; Hematologic response
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NICHE-AIHA: Patients who were diagnosed with AIHA in the investigating hospitals from Jan 1, 2001.
  Interventions: Other: A combined retrospective and prospective observational follow-up

INTERVENTIONS:
Other: A combined retrospective and prospective observational follow-up — The NICHE-AIHA will collect basic information, diagnostic and treatment information, as well as health costs information of patients from medical records. The study will use questionnaire to measure the exposure of patients, and prospectively follow-up to collect the prognosis information.

SUMMARY:
Hematological diseases are disorders of the blood and hematopoietic organs. The current hematological cohorts are mostly based on single-center or multi-center cases, or cohorts with limited sample size in China. There is a lack of comprehensive and large-scale prospective cohort studies in hematology.

The objectives of this study are to investigate the incidence and risk factors of autoimmune hemolytic anemia (AIHA) and to analyze the treatment effectiveness, patient prognosis and healthcare costs in China.

1. Analyze the demographic and clinical characteristics of patients with AIHA, including sex, age, disease severity, and other relevant factors.
2. Examine disease features of AIHA patients, such as biochemical and hematological indicators
3. Assess treatment patterns and real-world effectiveness in AIHA patients.
4. Evaluate clinical outcomes, including hematologic response, relapse, and mortality
5. Investigate long-term prognosis, including post-discontinuation outcomes and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with AIHA.
* Hemoglobin<100g/L
* Subjects treated at the Institute of Hematology and Blood Diseases Hospital from Jan 1, 2001.

Exclusion Criteria:

* Subject unlikely to be available for long-term follow-up for any reason (e.g., inability to obtain follow-up data or presence of severe comorbidities).
* Subject with alcohol or drug dependence may reduce their compliance with the study.
* Subjects that the investigator believes have other reasons that make them unsuitable for inclusion in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed as AIHA.
  Diagnostic criteria for AIHA (Autoimmune Hemolytic Anemia):
  Hemoglobin level meets the diagnostic threshold for anemia; Decreased serum haptoglobin (<250 mg/L), elevated total bilirubin (≥17.1 μmol/L, mainly indirect bilirubin), elevated lactate dehydrogenase (LDH), and reticulocyte percentage >4% or absolute reticulocyte count >120×10^9/L; Presence of autoantibodies against red blood cells.
Sampling Method: Non-Probability Sample
Enrollment: 9999 (Estimated)
Dates: Start 2001-01-01 (Actual); Primary Completion 2070-12-31 (Estimated); Study Completion 2070-12-31 (Estimated)

PRIMARY OUTCOMES:
Hematologic response | Assessments will be conducted at baseline, 6 months, 12 months, and 24 months after treatment, as well as at study completion, with an average interval of approximately 1 year.
  Hematologic response contains improvements in hemoglobin.

CONTACTS AND LOCATIONS:
Locations (1):
- Red Blood Cell Diseases Center and Regenerative Medicine Center, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No